CLINICAL TRIAL: NCT01245023
Title: Laparoscopic Adhesiolysis in Treatment of Chronic Abdominal Pain - a Prospective Randomized Trial
Brief Title: Adhesiolysis in Chronic Abdominal Pain
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: lack of funding
Sponsor: North Karelia Central Hospital (Other)
Responsible Party: Principal Investigator, Sanna Kouhia, MD, North Karelia Central Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NKCH-Surg-007
Record Dates: First submitted 2010-11-19; First posted 2010-11-22 (Estimated); Last update posted 2013-01-03 (Estimated); Status verified 2012-12

CONDITIONS: Chronic Abdominal Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- laparoscopy (Active Comparator): laparoscopic adhesiolysis and application of Sprayshield spray to prevent further adhesions
  Interventions: Procedure: Laparoscopic adhesiolysis
- placebo-control (Placebo Comparator): anaethesia and skin incisions without laparoscopy or related procedures
  Interventions: Procedure: Placebo-surgery

INTERVENTIONS:
Procedure: Laparoscopic adhesiolysis — Laparoscopic adhesiolysis and Sprayshield
  Arms: laparoscopy
Procedure: Placebo-surgery — skin incisions without laparoscopy or related procedures
  Arms: placebo-control

SUMMARY:
Laparoscopic adhesiolysis has been used in treatment of chronic abdominal pain. There has been only one previous controlled study, that stated laparoscopy alone had the same benefits than laparoscopic adhesiolysis. The aim of this study is to compare laparoscopic adhesiolysis with a placebo-procedure in chronic abdominal pain.

ELIGIBILITY:
Inclusion Criteria:

* age 18-65 years
* abdominal pain at least 6 months
* previous abdominal surgery and/or significant abdominal trauma and/or abdominal infection
* ASA class I-II

Exclusion Criteria:

* psychiatric disorder
* significant other somatic diseases (ASA class III-V)
* refusal to participate

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-01; Primary Completion 2016-12 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
pain | 6 months

CONTACTS AND LOCATIONS:
Locations (6):
- Finland (6):
  - Kainuu Central Hospital, Kajaani
  - Kuopio University Hospital, Kuopio
  - Mikkeli Central Hospital, Mikkeli
  - Oulu University Hospital, Oulu
  - Pieksämäki district hospital, Pieksämäki
  - Turku University Hospital, Turku